CLINICAL TRIAL: NCT00716612
Title: Effect of Coenzyme Q 10 Supplementation on Myalgia Induced by HMG-CoA Reductase Inhibitors
Brief Title: Does Coenzyme Q 10 Supplementation Reduce Muscle Pain Caused by Statins? (Cholesterol Lowering Medications)
Acronym: COSMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, David Rott, Consultant, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Solgar-080
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Statin Induced Myalgia
Keywords: Coenzyme Q 10; Statin; Myalgia
MeSH Terms: conditions — Myalgia | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): PO Placebo QD
  Interventions: Drug: Placebo control
- 1 (Experimental): PO Coenzyme Q 10 QD
  Interventions: Drug: Coenzyme Q 10

INTERVENTIONS:
Drug: Coenzyme Q 10 — PO Coenzyme Q 10 120 mg QD
  Other Names: ubiquinone
  Arms: 1
Drug: Placebo control — po Placebo QD
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Coenzyme Q 10 supplementation will decrease the rate of Muscle Pain in patients with previous statin related Muscle Pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for hyperlipidemia with a HMG-CoA reductase inhibitor (i.e. pravastatin, simvastatin rosuvastatin or atorvastatin) and reporting myopathic symptoms

Exclusion Criteria:

* Patients with other identifiable cause of myopathy. Patients with clinical evidence of hepatic, renal, or endocrine disease; coagulopathy; or other serious medical conditions will be excluded.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
1. The number of patients who tolerate statin at the initial dose. 2. The number of patients remaining on statin therapy. 3. Change in myalgia score. | 4, 8, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Rott, MD, Principal Investigator — Hadassah-Hebrew University Hospital
Locations (1):
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel